CLINICAL TRIAL: NCT04341493
Title: Treatment With Hydroxychloroquine vs Nitazoxanide + Hydroxychloroquine in Patients With COVID-19 With Risk Factors for Poor Outcome
Brief Title: Hydroxychloroquine vs Nitazoxanide in Patients With COVID-19
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Concerns about safety of Hydroxychloroquine
Sponsor: Hugo Mendieta Zeron (Other)
Responsible Party: Sponsor-Investigator, Hugo Mendieta Zeron, Chief of the Research Department, Materno-Perinatal Hospital of the State of Mexico
Organization: Materno-Perinatal Hospital of the State of Mexico (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-03-681
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus Infection
Keywords: Treatment; Evolution
MeSH Terms: conditions — Coronavirus Infections | interventions — nitazoxanide; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: In this study all patients with a COVID-19 positive result attended at the Health Institute of the State of Mexico (ISEM), will be invited to participate and offered one of two options that try to reduce the complications of this disease.
Who Masked: Participant
Masking Description: Patients won´t know whether the treatment they receive is hydroxychloroquine or nitazoxanide + hydroxychloroquine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide + hydroxychloroquine (Experimental): Hydroxychloroquine 400 mg PO every 12 hours for two days and then 200 mg PO every 12 hours for four days + Nitazoxanide 500 mg PO every 6 hours for six days
  Interventions: Drug: Nitazoxanide 500 MG; Drug: Hydroxychloroquine
- Hydroxychloroquine (Active Comparator): Hydroxychloroquine 200 mg PO every 12 hours for 7 days
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Nitazoxanide 500 MG — Clinical evaluation of patients with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) using this option with two drugs
  Other Names: hydroxychloroquine
  Arms: Nitazoxanide + hydroxychloroquine
Drug: Hydroxychloroquine — Clinical evaluation of patients with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) using this option with one drug

SUMMARY:
Coronaviruses (CoV) are positive-sense single-stranded RNA viruses that infect a wide range of hosts producing diseases ranging from the common cold to serious / fatal events. Nitazoxanide (NTZx) is a derivative of 5-nitrothiazole, synthesized in 1974 by Rosignol - Cavier. NTZx has powerful antiviral effects through the phosphorylation of protein kinase activated by double-stranded RNA, which leads to an increase in phosphorylated factor 2-alpha, an intracellular protein with antiviral effects. The purpose of this study is to contrast the beneficial effect of NTZx vs NTZx plus hydroxychloroquine in patients Coronavirus Disease (COVID-19) as well as against other treatments.

DETAILED DESCRIPTION:
Introduction The current pandemic caused by the SARS-COV2 coronavirus (COVID-19) is life-threatening and is challenging the world's best health systems. Accelerated spread of this pandemia led physicians to try a variety of treatments without a well established sequence due to ignorance about this new disease. The case fatality rate has been calculated at 2.2% but there are differences depending on the country affected.

Perspective When comparing the evolution of cases between Spain and Mexico, an apparently less pronounced trend is observed in Mexico, but this may be due to underdiagnosis. In calculations by the Mexican Ministry of Health, around 6% of the patients (approximately 10,500) who contract COVID-19 could be found serious and in need of hospitalization in intensive care.

NTZx NTZx and its circulating active metabolite, tizoxanide, inhibit the replication of a wide range of viruses, both RNA and DNA. It has action against 16 strains of Influenza A virus subtypes H1N1, H3N2, H3N2v, H3N8, H5N9, H7N1 and a strain of influenza B. It also works against respiratory syncytial virus, norovirus, dengue, yellow fever, Japanese encephalitis virus, rotavirus , hepatitis B and C, even against the human immunodeficiency virus (Severe Acute Respiratory Syndrome (SARS) and Middle East respiratory syndrome (MERS).

Problem Mexico is in Phase 2 according to the World Health Organization (WHO) and more local infections due to coronaviruses are expected. To date, various COVID-19 treatment schemes are being tested, but the usefulness of none can be assured.

When reviewing the drug schemes that are being carried out in the world, it calls the attention that developing countries are not included, beyond the fact that the tested alternatives are economically inaccessible.

This clinical survey aims to test the possible utility of NTZx against COVID-19, alone or in combination with hydroxychloroquine.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive patients
* Treated at the Health Institute of the State of Mexico (ISEM).
* With risk factors to get complicated: age more than 60 years old, diabetes mellitus or obesity grade II or more.

Exclusion Criteria:

* Patients who have inherent contraindications to each drug.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilation requirement | Since the diagnosis until two weeks after
  Percentage of patients COVID-19 positive that required mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: José Meneses Calderón, MD, Principal Investigator — Hospital Materno-Perinatal "Mónica Pretelini Sáenz"; Srivatsan Padmanabhan, MD, PhD, Principal Investigator — St. Joseph Medical Center
Locations (1):
- Materno-Perinatal Hospital "Mónica Pretelini", Toluca, Mexico

IPD SHARING:
Plan to Share IPD: Yes
If the final selected medical journal to send the paper of our research request it, we will add the full database of the studied population.
Supporting Information: Study Protocol, ICF
Time Frame: After finishing the study.
Access Criteria: Requested by the journal or after publication if any researcher in the world express interest if the information of this survey.

REFERENCES:
- [Background] Rossignol JF. Nitazoxanide, a new drug candidate for the treatment of Middle East respiratory syndrome coronavirus. J Infect Public Health. 2016 May-Jun;9(3):227-30. doi: 10.1016/j.jiph.2016.04.001. Epub 2016 Apr 16. PMID 27095301
- [Background] Mo Y, Fisher D. A review of treatment modalities for Middle East Respiratory Syndrome. J Antimicrob Chemother. 2016 Dec;71(12):3340-3350. doi: 10.1093/jac/dkw338. Epub 2016 Sep 1. PMID 27585965
- [Background] Li H, Wang YM, Xu JY, Cao B. [Potential antiviral therapeutics for 2019 Novel Coronavirus]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Mar 12;43(3):170-172. doi: 10.3760/cma.j.issn.1001-0939.2020.03.004. Chinese. PMID 32164080
- [Derived] Calderon JM, Zeron HM, Padmanabhan S. Treatment with Hydroxychloroquine vs Hydroxychloroquine + Nitazoxanide in COVID-19 patients with risk factors for poor prognosis: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jun 8;21(1):504. doi: 10.1186/s13063-020-04448-2. PMID 32513231